CLINICAL TRIAL: NCT01847287
Title: A Prospective, Observational, Single-blinded, Longitudinal Study of Natalizumab Effect on Brain Atrophy and Disability in Multiple Sclerosis Patients Over 5 Years.
Brief Title: A Longitudinal Study of Brain Atrophy in MS Patients Over 5 Years
Acronym: TST
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Director, Buffalo Neuroimaging Analysis Center, Professor, University at Buffalo
Other Study IDs: TST5
Record Dates: First submitted 2013-05-01; First posted 2013-05-06 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Tysabri; MRI; Natalizumab
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tysabri: All subjects took Tysabri and also had an MRI which we use for the baseline evaluation. Over 5 years, some patients remained on Tysabri, some started another drug and others were off Tysabri for a time but then restarted.

SUMMARY:
The primary aim of this study is to evaluate the effect of using Tysabri on changes in the brain using MRI and on disease progression in patients with relapsing-remitting Multiple Sclerosis over 5 years.

DETAILED DESCRIPTION:
This is a prospective, observational, single-blinded, longitudinal study of natalizumab effect on brain atrophy development and disability progression in multiple sclerosis patients over 5 years, which will evaluate originally treated patients with natalizumab who participated in a prospective 1- and 2-year VWMTR study. (Zivadinov et al., 2011b) All subjects will be assessed at 5-year follow-up with the same clinical examinations and will obtain 1.5T MRI examination on the same scanner that did not undergo any upgrade changes in the period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participation in natalizumab 1-year follow-up study
* Participants were aged 18-65
* Have clinically definite MS according to the Polman criteria of either RR or RSP disease type
* EDSS scores ≤6.5
* disease duration <30 years
* normal kidney function (creatinine clearance >59 mL/min)
* started therapy either with natalizumab or IM interferon beta-1a (IFNβ-1a)
* Signed informed consent
* Normal kidney functioning (creatinine clearance >59)
* None of the exclusion criteria

Exclusion Criteria:

* A clinically significant infectious illness (e.g., cellulitis, abscess, pneumonia, septicemia) within 30 days prior to 5-year follow-up visit
* Nursing mothers or pregnant women who will need to undergo 5-year follow-up MRI
* Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol
* Any other reasons that, in the opinion of the Investigator, indicate that the subject is unsuitable for enrollment into this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis - relapsing remitting
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The primary aim of this study is to define the effect of the number of natalizumab cycles on development of brain atrophy and progression of disability in originally treated patients with natalizumab in relapsing multiple sclerosis (MS). | 5 years
  Evaluation of MRI images from baseline in comparison with a 5 year MRI.

SECONDARY OUTCOMES:
The secondary objective of this study is to define the effect of the number of natalizumab cycles on accumulation of T2-LV and T1-LV and their VW-MTR changes over 5 years. | 5 years
  To evaluate any effect of the number of Tysabri cycles on lesion volume.

CONTACTS AND LOCATIONS:
Locations (1):
- Buffalo Neuroimaging Analysis Center, Buffalo, New York, United States